CLINICAL TRIAL: NCT04558957
Title: Prospective, Multi-centre Clinical Study to Assess the Safety and Efficacy of Mechanochemical Ablation With the Use of Flebogrif in Patients With Great Saphenous Vein Insufficiency
Brief Title: Clinical Study to Assess the Safety and Efficacy of Mechanochemical Ablation With Flebogrif in Patients With Great Saphenous Vein Insufficiency
Acronym: POLFLEB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balton Sp.zo.o. (Industry)
Collaborators: KCRI (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POLFLEB
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Chronic Venous Insufficiency, CVI
MeSH Terms: conditions — Blindness, Cortical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FLEBOGRIF (Experimental): Interventions will be performed using Flebogrif catheter.
  Interventions: Device: FLEBOGRIF

INTERVENTIONS:
Device: FLEBOGRIF — The catheter is a device dedicated to mechano-chemical ablation of insufficient veins of the superficial system.

SUMMARY:
The objective of the study is to collect clinical data of patients in whom Flebogrif® will have been used for mechanochemical ablation of incompetent veins in the follow-up period, as related to the safety, clinical effectiveness, properties and advantages of Flebogrif®.

The proposed study is a prospective, multi-centre clinical trial assessing the safety, efficacy and quality of Flebogrif® in a population of patients with the incompetent great saphenous vein, who require surgical treatment.

ELIGIBILITY:
Study inclusion criteria:

1. Signing the Informed Consent Form by the patient found eligible for the treatment with the mechanochemical method
2. The patient declares willingness to participate in the study and in the monitoring visits envisaged in the study protocol
3. A patient with diagnosed varicose veins and diagnosed great saphenous vein (GSV) insufficiency confirmed by ultrasound (CEAP class C2-C6)
4. Favourable anatomy enabling the introduction of the Flebogrif® guidewire/catheter and positioning of its top part at the dedicated site (2-3 cm below SFJ)
5. Diameter of the treated vein of 4-10 mm
6. No data or no history indicating an allergy to the sclerosing chemicals used in the mechanochemical method (polidocanol), on the basis of the information obtained from the patient and the available medical records
7. No clinical symptoms indicating (chronic, critical) lower limb ischaemia precluding the use of compression, on the basis of a physical examination or, in unclear cases, of a Doppler ultrasound examination
8. No medical information or no history of coagulation system dysfunction of the type of thrombophilia or bleeding diatheses
9. No cutaneous lesions (purulent, bullous) within the limb found eligible for treatment with the mechanochemical method
10. No clinical data indicating recent thrombosis within the deep vein system
11. No clinical data on diabetes with vascular complications
12. No clinical data indicating an active neoplastic process

Study exclusion criteria:

1. Recent deep vein thrombosis or occlusion
2. Congenital disorders with associated occlusion of deep system veins
3. Pregnancy and breast-feeding
4. Lower limb ischaemia
5. Severe lymphatic oedema
6. Bleeding diatheses
7. Documented allergic reaction to sclerosing chemicals used in mechanochemical vein ablation
8. Purulent dermatoses affecting the limb found eligible for treatment with mechanochemical vein ablation
9. Previous procedures on insufficiency veins of the superficial system
10. Acute infection
11. History of great saphenous vein thrombosis
12. End-stage kidney disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Primary efficacy endpoint: Occlusion rate | 3 months
  Primary efficacy endpoint: Occlusion rate of the great saphenous vein in the treated segment at 3 months
Primary safety endpoint: Rate of SAE | 30 days after the procedure
  Primary safety endpoint: Rate of serious adverse events within 30 days after the procedure

SECONDARY OUTCOMES:
Occlusion rate | 1, 6, 12, 18, 24 months
  Occlusion rate of the great saphenous vein at 1, 6, 12, 18 and 24 months
Number of Participants with no reflux in treated segment of the vein | 1, 3, 6, 12, 18, 24 months
  Number of Participants with no reflux in the treated segment of the great saphenous vein at 1, 3, 6, 12, 18 and 24 months
Change in quality of life by Aberdeen Varicose Vein Questionnaire | 12 and 24 months
  Change in quality of life measured with the use of the Aberdeen Varicose Vein Questionnaire at 12 and 24 months
  Scale score: 0-100; higher score = worse outcome.
Clinical success - changes in rVCSS | 12 and 24 months
  Clinical success, defined as change in rVCSS classification (Revised Venous Clinical Severity Score) after 12 and 24 months
  Scale score 0-30; higher score = worse outcome.
Assessment of pain during the procedure | During procedure
  Assessment of pain during the procedure (Visual Analogue Pain Scale, VAPS) ranging from 0 to 10. Pain assessed using the Visual Analogue Scale (range 0-10; 0 = no pain; 2 = mild pain, 4 = nagging, annoying pain; 6 = severe pain; 8 = very severe pain; 10 = unbearable pain).
Assessment of pain within 0-7 days after the procedure: Visual Analogue Scale | 0-7 days after procedure
  Assessment of pain within 0-7 days after the procedure (VAPS 0-10, daily assessment). Pain assessed using the Visual Analogue Scale (range 0-10; 0 = no pain; 2 = mild pain, 4 = nagging, annoying pain; 6 = severe pain; 8 = very severe pain; 10 = unbearable pain).
Assessment of the need for analgesic treatment | 0-7 days after procedure
  Assessment of the need for analgesic treatment after the procedure (0-7 days)
Period needed to resume normal activities | up to 2 years after the treatment
  Period needed to resume normal activities
Period needed to return to work (sick leave period) | up to 2 years after the treatment
  Period needed to return to work (sick leave period)
Complications rate | up to 2 years after the treatment
  Complications rate including deep vein thrombosis, nerve damage, infections, etc.

CONTACTS AND LOCATIONS:
Locations (4):
- Poland (4):
  - Centrum Chirurgii i Stomatologii Jaworuccy Sp. P., Gorzów Wielkopolski
  - Centrum Medyczne Angelius Provita; Europejskie Centrum Flebologii, Katowice
  - Medyczne Centrum Nałęczów sp. z o.o., Lublin
  - Klinika Dorobisz, Wroclaw